CLINICAL TRIAL: NCT04136132
Title: Establishment of a Monocentric and Prospective Clinico-biological Database in Patients With Pancreatic Adenocarcinoma
Brief Title: Prospective Monocentric Clinical-biological Database
Acronym: BCBPancréas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PROICM 2018-10 BPA
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Cancer
Keywords: oncology; Pancreatic
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological collection (Experimental): Biological collection
  For all the patients include in the study :
  blood and tissue samples collected before and during treatment. In parallel to this biological collection, standardized clinical data will be entered into a database
  Interventions: Other: Biological collection

INTERVENTIONS:
Other: Biological collection — The biological collection will also include samples of blood samples collected before or after surgery but also samples frozen and/or paraffin-embedded tissue sections.

SUMMARY:
Pancreatic adenocarcinoma (PA) is a solid cancer with a very poor prognosis with overall survival, all stages combined, not exceeding 5% at 5 years. The incidence and number of deaths caused by this type of tumor have been steadily increasing for two decades. In the absence of therapeutic advances, PA will be one of the leading causes of cancer deaths in 2030.

In recent years, researchers and clinicians have now attempted to characterize and understand PA as a whole, through the various stages of its carcinogenesis and the analysis of its microenvironment. Indeed, the stroma of PA can represent up to 80% of the tumor mass and mainly composed of activated fibroblasts (CAF), endothelial and immune cells and extracellular matrix (collagen and fibronectin). However, the characterization of cell subtypes of this stroma is under study, as the pro or anti-tumor role of each cell subtype is not yet well understood.

New technologies such as the CyTOF that has just been acquired by the ICM and the IRCM will make it possible to study these problems and to examine the cellular subpopulations that make up the tumor. On the other hand, active research is conducted to disrupt the dialogue between the tumor cells and those of the microenvironment.

The search for innovative treatments in pancreatic adenocarcinoma requires the use of models of relevant preclinical studies. The most widely used models are based on cell lines of human origin used in vitro or in vivo after xenograft in immunodeficient mice. In particular, studies with pancreatic adenocarcinomas (PDX) derived tumors of patients reported that the response rate of PDX to certain drugs (gemcitabine, erlotinib ...) used clinically was similar to the response rates of patients enrolled in clinical studies. of these agents as monotherapy. A number of studies have evaluated the efficacy of targeted anti-tumor, anti-angiogenic or anti-stroma therapies from these PDTX models. Personalized medicine strategies can be envisioned as well as the study of new biomarkers, drugs or molecular mechanisms involved in therapeutic resistance. For several years, the investigators have been developing AP PTDX in the INSERM 1194 unit.

The investigators propose to continue the development of this collection of pancreatic adenocarcinoma PDTX prospectively and to carry out their histological, molecular and mutational characterization.

DETAILED DESCRIPTION:
Pancreatic adenocarcinoma (PA) is a solid cancer with a very poor prognosis with overall survival, all stages combined, not exceeding 5% at 5 years. The incidence and number of deaths caused by this type of tumor have been steadily increasing for two decades. In the absence of therapeutic advances, AP will be one of the leading causes of cancer deaths in 2030. The poor prognosis of PA is explained by a diagnosis often late and by the biological characteristics of the tumor, marked by significant heterogeneity, hypovascularization and an abundant desmoplastic stroma explaining resistance to different treatments. PA results from the successive accumulation of genetic and epigenetic alterations (mutations, hypermethylation, overexpression) marking the transformation of the pancreatic epithelium into localized adenocarcinoma and then rapidly metastatic. Surgery, the only potentially curative treatment, is only possible for 5 to 10% of patients. For these resectable tumors, only 20% of fully operated patients are alive at 5 years. At the metastatic stage, chemotherapies, used in combination with symptomatic treatments, have limited efficacy. The standard treatments are gemcitabine and in recent years, FOLFIRINOX (5-FU combination, irinotecan and oxaliplatin), the effectiveness of which is associated with significant toxicities that limit its administration to patients with preserved general condition (Conroy, 2011). Recently, the Nab-Paclitaxel (albumin-based paclitaxel) has shown an interesting efficiency but is still not accessible outside of clinical studies. Despite these advances, the results remain modest, with overall patient survival increased by 6 months on gemcitabine, 11 months on FOLFIRINOX and 8.5 months on GEMBRAX (gemcitabine + Nab-Paclitaxel. Thus, oncologists lack solutions. Therapeutics after Progression to the First Line of Chemotherapy Many clinical trials have attempted to combine other chemotherapies or targeted therapies with relatively low survival gains.

In preclinical studies, the search for new therapies initially focused on the pancreatic cancer cell by targeting the affected proteins and signaling pathways and then the microenvironment was identified as a potential target. Various inhibitors have been considered to target the MEK1 / 2, PI3K-mTOR, JAK-STAT and Notch pathways with often disappointing clinical results. Other preclinical work requires further studies, such as those targeting the CXCR4, TGFb or PARP pathways. Targeting of tyrosine kinase receptors has been widely studied but remains relevant with a number of ongoing studies using inhibitors of EGFR, IGFR or cMET family members.

In recent years, researchers and clinicians have now attempted to characterize and understand PA as a whole, through the various stages of its carcinogenesis and the analysis of its microenvironment. Indeed, the stroma of PA can represent up to 80% of the tumor mass and mainly composed of activated fibroblasts (CAF), endothelial and immune cells and extracellular matrix (collagen and fibronectin). It is in this sense that research is now evolving by identifying targets and interactions at the stroma level. Therapeutic trials including SHH inhibitors (Saridegib), hyaluronidases to destroy extracellular matrix (PEGPH20), inhibitors of RTK or their ligands (FGFR, VEGFR, PDGFR), or sensitive alkylating agents only under hypoxic conditions (1). evofosfamide (TH-302)) were studied. By inhibiting this microenvironment, the goal is also to increase the penetration of drugs within the tumor. However, the characterization of cell subtypes of this stroma is under study, as the pro or anti-tumor role of each cell subtype is not yet well understood. New technologies such as the CyTOF that has just been acquired by the ICM and the IRCM will make it possible to study these problems and to examine the cellular subpopulations that make up the tumor. On the other hand, active research is conducted to disrupt the dialogue between the tumor cells and those of the microenvironment. Indeed the stroma is a secretory environment (and particularly via activated fibroblasts (CAF)), in constant interaction with the tumor cells, which themselves secrete factors that will activate the fibroblasts. It is in this context that part of the preclinical research conducted at the IRCM aims to target this dialogue and inhibit pro-tumor CAF.

Finally, immune cells are a major component of this stroma, although in pancreatic cancer the microenvironment is highly immunosuppressive, associated with low lymphocyte infiltration and increased macrophage-type 2 infiltration, MDSCs, and lymphocytes. T regulators. Current results using anti-immune "checkpoint" antibodies are controversial, but the activation of the immune system in this pathology nevertheless remains totally relevant.

Pre-clinical model of AP The search for innovative treatments in pancreatic adenocarcinoma requires the use of models of relevant preclinical studies. The most widely used models are based on cell lines of human origin used in vitro or in vivo after xenograft in immunodeficient mice. Nevertheless, these models are based on a limited number of lines, largely selected by performing cell cultures in vitro before their implantation in animals. They therefore do not reflect the characteristics of human tumors or their biological heterogeneity and do not include a representation of the microenvironment nor the peritumoral stroma, which nevertheless plays a major role in the progression of the disease. In parallel with cell lines, transgenic mouse models have been developed and have become essential for studying the carcinogenesis of PA. These models, although artificial, remain very interesting for the fundamental study of pancreatic carcinogenesis (tumor cells and microenvironment) and the test of non-targeted therapies that can act on murine cells. However, they remain limited to test new targeted treatments specific to human proteins. In addition, the low incidence of the adenocarcinoma stage and the window of time between the onset of AP and the death of the mouse (a few weeks) remains problematic for the implementation of therapeutic protocols.

Patient-derived tumors (PTDX) represent another type of promising study model. These PTDX are established from small tumor fragments obtained during surgical operations of patients with AP and grafted directly and then successively to immunodeficient mice until their stabilization. The development of a significant collection of PA xenografts directly transplanted to the nude mouse and their conservation represents one of the current solutions for obtaining preclinical models as close as possible to the tumors encountered in the clinic. Subsequently kept frozen, they can be used as a reliable model because they retain the histological and molecular characteristics of the source tumors. The major disadvantage is the use of immunocompromised animals in which all immune cells are not active so the role of immunity may be only partially studied. The characteristics of the tumor (genotype, phenotype, structure) and the cellular heterogeneity seem to be preserved during the passages and to stabilize at the passage 3. The human stroma is however progressively replaced by the stroma of the mouse. In particular, studies with pancreatic adenocarcinoma PDXs have reported that the response rate of PDX to certain drugs (gemcitabine, erlotinib ...) used clinically is similar to the response rates of patients enrolled in clinical studies of these agents as monotherapy. A number of studies have evaluated the efficacy of targeted anti-tumor, anti-angiogenic or anti-stroma therapies from these PDTX models. Personalized medicine strategies can be envisioned as well as the study of new biomarkers, drugs or molecular mechanisms involved in therapeutic resistance. For several years, the investigators have been developing AP PTDX in the INSERM 1194 unit, some of which are in the process of being characterized and are the basis of several translational research projects on the IRCM website (Targeting study receptors of the TAM family ; Inhibition of the dialogue between CAF and tumor cells; Study of resistance to gemcitabine and Folfirinox.

ELIGIBILITY:
Inclusion Criteria:

* Patient over the age of 18;
* Patient managed for pancreatic adenocarcinoma;
* Patient eligible for at least one (or more) surgery (s) and chemotherapy;
* Patient giving informed consent

Exclusion Criteria:

* Patient not affiliated to a social security scheme;
* Pregnant and / or nursing patient;
* Patient under guardianship, curatorship or safeguard of justice;
* Patient whose regular follow-up is impossible for psychological, family, social or geographical reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2034-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who gave their consent to participate in the study | Until the study completion: 8 years
  The proportion of patients who consent to participate in the study among the screened patients

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Emmanuel COLOMBO, MD, Study Chair — Institut Régional du Cancer de Montpellier (ICM)
Locations (1):
- Institut Régional du Cancer de Montpellier, Montpellier, Occ, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rahib L, Smith BD, Aizenberg R, Rosenzweig AB, Fleshman JM, Matrisian LM. Projecting cancer incidence and deaths to 2030: the unexpected burden of thyroid, liver, and pancreas cancers in the United States. Cancer Res. 2014 Jun 1;74(11):2913-21. doi: 10.1158/0008-5472.CAN-14-0155. PMID 24840647
- [Background] Garrido-Laguna I, Hidalgo M. Pancreatic cancer: from state-of-the-art treatments to promising novel therapies. Nat Rev Clin Oncol. 2015 Jun;12(6):319-34. doi: 10.1038/nrclinonc.2015.53. Epub 2015 Mar 31. PMID 25824606
- [Background] Chiorean EG, Coveler AL. Pancreatic cancer: optimizing treatment options, new, and emerging targeted therapies. Drug Des Devel Ther. 2015 Jul 7;9:3529-45. doi: 10.2147/DDDT.S60328. eCollection 2015. PMID 26185420
- [Background] Rubio-Viqueira B, Jimeno A, Cusatis G, Zhang X, Iacobuzio-Donahue C, Karikari C, Shi C, Danenberg K, Danenberg PV, Kuramochi H, Tanaka K, Singh S, Salimi-Moosavi H, Bouraoud N, Amador ML, Altiok S, Kulesza P, Yeo C, Messersmith W, Eshleman J, Hruban RH, Maitra A, Hidalgo M. An in vivo platform for translational drug development in pancreatic cancer. Clin Cancer Res. 2006 Aug 1;12(15):4652-61. doi: 10.1158/1078-0432.CCR-06-0113. PMID 16899615
- [Background] Leconet W, Larbouret C, Chardes T, Thomas G, Neiveyans M, Busson M, Jarlier M, Radosevic-Robin N, Pugniere M, Bernex F, Penault-Llorca F, Pasquet JM, Pelegrin A, Robert B. Preclinical validation of AXL receptor as a target for antibody-based pancreatic cancer immunotherapy. Oncogene. 2014 Nov 20;33(47):5405-14. doi: 10.1038/onc.2013.487. Epub 2013 Nov 18. PMID 24240689
- [Background] Ogier C, Colombo PE, Bousquet C, Canterel-Thouennon L, Sicard P, Garambois V, Thomas G, Gaborit N, Jarlier M, Pirot N, Pugniere M, Vie N, Gongora C, Martineau P, Robert B, Pelegrin A, Chardes T, Larbouret C. Targeting the NRG1/HER3 pathway in tumor cells and cancer-associated fibroblasts with an anti-neuregulin 1 antibody inhibits tumor growth in pre-clinical models of pancreatic cancer. Cancer Lett. 2018 Sep 28;432:227-236. doi: 10.1016/j.canlet.2018.06.023. Epub 2018 Jun 20. PMID 29935372